CLINICAL TRIAL: NCT06616259
Title: First-line Treatment of MCapOX in Combination with Cetuximab Versus MFOLFOX6 in Combination with Cetuximab for RAS/BRAF Wild-type, MSS, Unresectable Left-Sided Metastatic Colorectal Cancer: a Multicenter, Randomized, Controlled, Phase III Study
Brief Title: First-line Treatment of MCapOX + Cetuximab Vs. MFOLFOX6 + Cetuximab for RAS/BRAF Wild-type, MSS, Unresectable Left-Sided MCRC: a Multicenter, Randomized, Controlled, Phase III Study
Acronym: CAPCET-III
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Meng Qiu (Other)
Responsible Party: Sponsor-Investigator, Meng Qiu, Principal Investigator, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240716
Record Dates: First submitted 2024-09-17; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer (CRC); Capecitabine; Cetuximab
Keywords: CAPCET-III
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): mCapOX (Capecitabine+Oxaliplatin) plus Cetuximab
  Interventions: Drug: mCapOX plus Cetuximab
- Arm B (Active Comparator): mFOLFOX6 (Fluorouracil+Leucovorin+Oxaliplatin) plus Cetuximab
  Interventions: Drug: mFOLFOX6 plus Cetuximab

INTERVENTIONS:
Drug: mCapOX plus Cetuximab — mCapOX plus Cetuximab Induction therapy：Capecitabine 1000mg/m2 po, bid, D1-7 + Oxaliplatin ivgtt 85mg/m2, D1 + Cetuximab ivgtt 500mg/m2, D1; Q2W. Up to 12 cycle, if no progression, enter maintenance therapy.
  Maintenance therapy: Capecitabine 1000mg/m2 po, bid, D1-7 + Cetuximab ivgtt 500mg/m2, D1; Q2W. Until disease progression or toxicity is not tolerated. Cetuximab can be discontinued alone if not tolerated.
  Treatment after progression of maintenance therapy: Participants have the option to accept reintroducing the first-line induction chemotherapy regimen (mCapOx or mFOLFOX6 in combination with cetuximab) or accept second-line therapy.
  Arms: Arm A
Drug: mFOLFOX6 plus Cetuximab — mFOLFOX6 plus Cetuximab Induction therapy：Oxaliplatin ivgtt 85mg/m2, D1 + Leucovorin ivgtt 400mg/m2, D1 + Fluorouracil iv bolus 400mg/m2, D1 + Fluorouracil 2400mg/m2 continuous infusion for 46-48h + Cetuximab ivgtt 500mg/m2, D1; Q2W. Up to 12 cycle, if no progression, enter maintenance therapy.
  Maintenance therapy: Capecitabine 1000mg/m2 po, bid, D1-7 + Cetuximab ivgtt 500mg/m2, D1; Q2W. Until disease progression or toxicity is not tolerated. Cetuximab can be discontinued alone if not tolerated.
  Treatment after progression of maintenance therapy: Participants have the option to accept reintroducing the first-line induction chemotherapy regimen (mCapOx or mFOLFOX6 in combination with cetuximab) or accept second-line therapy.
  Arms: Arm B

SUMMARY:
This multicenter, randomized, controlled, phase III study is conducted to evaluate the efficacy and safety of first line mCapOX plus Cetuximab versus mFOLFOX6 plus Cetuximab for RAS/BRAF wild-type, MSS, Unresectable Left-Sided mCRC.

DETAILED DESCRIPTION:
Study participants who meet the enrollment criteria will be randomly assigned in a 1:1 ratio to either the mCapOX + cetuximab or mFOLFOX6 + cetuximab treatment groups, and those who have achieved control of their disease (Complete response [CR] + Partial response [PR] + Stable disease [SD]) after a maximum of 12 cycles of first-line induction therapy in both groups will continue to receive Capecitabine or Capecitabine + Cetuximab maintenance therapy until disease progression or toxicity is not tolerated or informed consent is withdrawn.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent and can understand and comply with the requirements of the study.
* Men and women ≥ 18 years of age.
* Patients with histologically or cytologically confirmed RAS and BRAF wild-type, MSS/pMMR, metastatic left-sided colorectal adenocarcinoma.
* Presence of at least one evaluable lesion, as defined in RECIST Version 1.1.
* With an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* No palliative first-line chemotherapy, targeted, immunotherapy, or prior platinum-based adjuvant chemotherapy, relapse more than 12 months from the end of adjuvant chemotherapy.
* According to the imaging findings and surgical assessment of initial unresectable, synchronous metastatic colorectal cancer, no serious complications of the primary tumor (obstruction, perforation, massive hemorrhage that cannot be treated in internal medicine, etc.) .
* Requirements for lab indicators: neutrophils ≥ 1.5 × 10^9/L, platelets ≥ 75 × 10^9/L, hemoglobin ≥ 8 g/dL; total bilirubin ≤ 1.5 × upper limit of normal (UNL); ASAT (SGOT) and/or ALAT (SGPT) ≤ 2.5 × UNL (≤ 5 × UNL if liver metastases); alkaline phosphatase ≤ 2.5 × UNL (≤ 5 × UNL if liver metastases, ≤ 10 × UNL if bone metastases); LDH < 1500 U/L; creatinine clearance (calculated according to Cockcroft and Gault formula) > 50 mL/min or serum creatinine ≤ 1.5 × UNL.

Exclusion Criteria:

* Patients with mCRC who were initially resectable with R0 resection or radiofrequency or SBRT were excluded.
* Patients diagnosed with MSI-H or dMMR by PCR or immunohistochemistry
* Hypersensitivity to any therapeutic agent.
* Patients who received adjuvant chemotherapy containing oxaliplatin and fluorouracil within 12 months before entering the study.
* Patients who have failed one or more palliative chemotherapy regimens.
* Patients with uncontrolled hepatitis B virus.
* Peripheral neuropathy ≥ CTC grade 2.
* Neurological or psychiatric disorders affecting cognitive performance.
* Patients with central nervous system metastasis could not be controlled with radiotherapy.
* Previous enteritis, chronic diarrhea, or recurrent bowel obstruction; uncontrolled bleeding from internal medicine; bowel perforation.
* Uncontrolled concomitant diseases within 6 months before the study, including unstable angina, acute myocardial infarction, cerebrovascular accident, etc.
* Pregnant or lactating patients, or those of childbearing potential who do not take adequate contraceptive measures.
* History of other malignancies, but no disease-free survival longer than 5 years.
* Patients concurrently receiving other anti-tumor treatment or participating in other interventional clinical trials.
* Patients who are unable to comply with this study for psychological, family or social reasons.
* Patients with other serious diseases that the investigator considers not suitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Estimated)
Dates: Start 2024-09-26 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | up to 3 years
  Progression free survival is defined as the period from randomization to disease progress or death. Includes first-line induction therapy and maintenance therapy.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 6 months
  Defined as the proportion of participants acquired Complete response (CR) or Partial response (PR) during treatment. Based on RECIST 1.1.
Disease control rate (DCR) | 6 months
  Defined as the proportion of patients who acquired Complete response (CR), Partial response (PR), or Stable disease (SD) during treatment. Based on RECIST 1.1.
Time to Failure of Strategy (TFS) | up to 3 years
  Defined as the time from the date of randomization to [secondary disease progression after reintroduction of first-line induction chemotherapy following maintenance therapy disease progression] or [all-cause death].
  If participants progressed on maintenance therapy after first-line induction chemotherapy without reintroduction of first-line induction chemotherapy or progressed during first-line induction chemotherapy, TFS equals PFS
Overall Survival (OS) | up to 5 years
  Defined as the period from randomization to death from any cause
Adverse Event rate | up to 3 years
  The rate of adverse event after treatment
Pharmacoeconomic | up to 3 years
  Including CERs (Cost-Effectiveness Ratios) and ICERs (Incremental Cost-Effectiveness Ratios).
  CERs：Defined as the ratio of the total costs of a medical intervention to the health benefits gained from that intervention.
  ICERs：Defined as the ratio of the difference in costs between two alternative interventions（Arm A and Arm B） to the difference in their effectiveness.
Quality of Life | up to 3 years
  Assessment of quality of life through the Quality of Life Questionnaire (QLQ)

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No